CLINICAL TRIAL: NCT04969081
Title: Augmenting Early Phase Substance Use Treatment With Therapeutic Work Activity to Improve Clinical Outcomes: a New Indication for an Old Intervention
Brief Title: Impact of Work Activity on SUD Outcomes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D3493-R
Record Dates: First submitted 2021-07-01; First posted 2021-07-20 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Substance-related Disorders
Keywords: substance-related disorders; rehabilitation, vocational
MeSH Terms: conditions — Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Two branch study: one branch for Vets not interested in competitive employment, and one for Vets interested in competitive employment. Within each branch, Veterans will be randomized to either treatment as usual, or treatment as usual plus referral to competitive or non-competitive work-focused program.
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blind to randomization status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment as usual (Active Comparator): usual substance use treatment
  Interventions: Other: treatment as usual
- treatment as usual plus referral to work focused program (Experimental): usual substance use treatment plus referral to a competitive or non-competitive work-focused program
  Interventions: Behavioral: referral to work focused program; Other: treatment as usual

INTERVENTIONS:
Behavioral: referral to work focused program — referral to Incentive Therapy or to Other Therapeutic and Supported Employment Services
  Arms: treatment as usual plus referral to work focused program
Other: treatment as usual — usual treatment

SUMMARY:
To date, there are no studies of the therapeutic effects of varied work-focused programs in Veterans undergoing outpatient substance use disorder (SUD) treatment. The investigators propose a randomized clinical trial to test the effects of work-focused programs on improving sobriety and other clinical outcomes in Veterans early in the course of recovery from SUD. Veterans will be randomized to either receive or not receive referral for work-focused therapeutic programs. Primary aim is to examine effects of work-focused programs on sobriety outcomes, namely sobriety and global functioning. Secondary aim is to examine effects of work-focused programs on psychiatric symptoms, self esteem/efficacy, and quality of life.

DETAILED DESCRIPTION:
The investigators propose a trial to test the effects of Incentive Therapy (IT) and Other Therapeutic and Supported Employment Services (Other TSES) on improving SUD outcomes in newly recovering Veterans in outpatient treatment. In line with eligibility criteria for different TSES programs, the investigators will employ a two branch study: One branch will be for Veterans who are not interested in pursuing competitive employment, and will be a two arm RCT with randomization (2:1) to referral for IT + treatment as usual (TAU; including usual SUD outpatient treatment) or TAU alone. The second branch will be for Veterans who express interest in competitive employment, and will be a two arm RCT with randomization (2:1) to referral for TSES competitive employment services + TAU or TAU alone. Total Intent to Treat sample will be 140 (n=70 per branch). Primary outcomes will be percent days abstinent during 3 month active phase and clinical global impression scale scores at 6 months. Secondary outcome will be psychiatric symptoms, self esteem/efficacy and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be Veterans enrolled in VACHS substance use treatment, who at time of consenting into the study are within 30 days of detoxification or last substance use as per medical record.
* Additional criteria will be as follows:

  * 18 years of age and older,
  * meeting DSM-V criteria for any current Substance Use Disorder (SUD) (e.g., opioids, cocaine, marijuana, amphetamine, or alcohol),
  * competent to give written informed consent and HIPAA authorization.

Exclusion Criteria:

* involvement in a legal case that may lead to incarceration during study period;
* developmental disability or medical illness that would prevent therapeutic work activity, as judged by PI or clinical staff providing this service;
* plans to relocate outside geographic area that would make follow-up unlikely;
* and/or lack of willingness to provide contact information of someone who can help us contact the participant in the event that we are unable to maintain contact directly.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
percent days abstinent | 3 months
  percent days abstinent during 3-month active phase
Clinical Global Impression | 6 months
  Clinical Global Impression ratings conducted at 6 months from study entry.

SECONDARY OUTCOMES:
change from baseline in BASIS-24 | 3 months
  change in Behavior and Symptom Identification Scale, self-report
change from baseline in Rosenberg self-esteem scale | 6 months
  change in self report of self-esteem
change from baseline in New General Self-Efficacy Scale | 6 months
  change in self-report of self-efficacy
change in WHOQOL BREF | 6 months
  change in self-report of quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Joanna M. Fiszdon, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified, anonymized dataset will be created. This dataset may be shared with other investigators, upon written request, under a data use agreement prohibiting the recipient from identifying or re-de-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset. The data sharing agreement will also restrict redistribution to third parties and proper acknowledgment of the data source. These datasets will be shared per guidelines provided by VACHS Information Security Officer.
Supporting Information: Study Protocol, SAP
Time Frame: After study completion
Access Criteria: After study completion for no less than 7 years.

DOCUMENTS (1):
  • Informed Consent Form (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT04969081/ICF_000.pdf